CLINICAL TRIAL: NCT03165136
Title: Prévention Des Fausses Couches Spontanées Répétées Par Hydroxychloroquine. Essai thérapeutique Multicentrique, randomisé, en Double Insu, Contre Placebo
Brief Title: Hydroxychloroquine for Prevention of Recurrent Miscarriage.
Acronym: BBQ
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29BRC16.0045
Record Dates: First submitted 2017-05-03; First posted 2017-05-24 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Miscarriage; First Trimester Abortion
Keywords: Unexplained Recurrent Miscarriage; First trimester abortion; Hydroxychloroquine; Antiphospholipid antibody
MeSH Terms: conditions — Abortion, Habitual | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Double Blind Randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active drug and placebo will be exactly the same
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental): The treatment will be orally administrated, at a daily dose of 400 mg of hydroxychloroquine . The treatment will be started before conception and will be stopped at the end of the tenth week of gestation or before in case of pregnancy loss.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): A similar placebo will be orally administrated every day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine : 200 mg twice a day
  Arms: Hydroxychloroquine
Drug: Placebo — placebo of hydroxychloroquine
  Arms: Placebo

SUMMARY:
Recurrent miscarriage (RM) defined by >=3 consecutive losses affects 1% of fertile couples. Most women have recurrent early loss with a failure of development before 10 weeks' gestation. Standard investigations fail to reveal any apparent cause in >50% of couples.

No study has demonstrated any benefit of any medication in women with Unexplained RM, in the presence or absence of an inherited thrombophilia.

Moreover, the benefit of aspirin and/or heparin has not been proved in women with Antiphospholipid (APL) antibody without other clinical manifestations of Antiphospholipid Syndrome.

Hydroxychloroquine (HQ) is a molecule whose properties (anti-thrombotic, vascular-protective, immunomodulatory, improved glucose tolerance, lipid-lowering, anti-infectious) could be useful against mechanisms of Unexplained RM.

There is no data concerning the benefit of HQ in RM in the presence or absence of antiphospholipid antibodies or any inherited thrombophilia.

Administration in (Systemic Lupus erythematosus (SLE) women and for Malaria prevention provides extensive safety data during pregnancy.

Oral administration makes possible treatment since the preconception period. For all of that and its low cost, hydroxychloroquine should be evaluated in RM whatever the woman thrombophilic status.

DETAILED DESCRIPTION:
Regarding the mechanisms of unexplained RM, on the basis of animal models and clinical studies, many hypotheses were raised:

* Reduced ovarian reserve,
* Progesterone defect: a double-blind trial did not show any benefit of progesterone therapy.
* Thrombotic mechanisms and/or endothelial dysfunction: An association with some inherited thrombophilias was suggested. A prothrombotic state outside of pregnancy was measured in women with previous RM and without known thrombophilia.
* Immunological disturbances (high titers of anti-thyroid or APL antibodies, maternal carriage of specific HLA alleles and immunological reactions against male-specific minor antigens, increased numbers of peripheral blood natural killer, overexpression of TOLL receptors, increase of TH1 and TH17 processes). Consequently, immunomodulatory treatments were proposed and assessed (no impact of intravenous immunoglobulins and no conclusive benefit of corticosteroids).
* Miscellaneous: BMI> 30 and chronic endometritis. Besides, the experience gained from previous clinical trials in RM leads us to emphasize, that subcutaneous administration of heparin limits its assessment among fertile women. Indeed, the treatment could not be administrated before conception and consequently the exposure was often too short (injections cannot be routinely initiated before 5 weeks).

Except psychological support, there is no treatment whose benefit has been proved in unexplained RM, in the presence or in the absence of an inherited thrombophilia. Moreover the absence of benefit of some treatments has been clearly demonstrated. Although the prognostic is not so poor (live-birth rates around 70%), proposed therapeutic interventions are sometimes excessive (regarding possible side effects and cost): as intravenous immunoglobulins, assisted procreation ...anti-TNF.

Consequently, for the management of these distressed patients, investigating other therapeutic options is highly needed.

Regarding recurrent miscarriage in women with high titers of antiphospholipid but without any other previous clinical event listed in the antiphospholipid syndrome, the benefit of antithrombotic treatment remains controversial (negative results of the HepASA trial) and hydroxychloroquine has never been assessed, although retrospective studies are encouraging.

ELIGIBILITY:
Inclusion Criteria:

* women aged from 18 to 38 years,
* women trying to conceive,
* women with at least 3 previous consecutive miscarriage in the first pregnancy trimester, of unknown origin (normal parental karyotypes, no uterine cavity abnormality, no antiphospholipid syndrome with other clinical events than RM in the first trimester of pregnancy.)
* women who have given their informed consent

Exclusion Criteria:

* ongoing pregnancy,
* Normal pregnancy since the last miscarriage,
* Uterine cavity abnormality,
* Abnormal parental karyotype,
* Antiphospholipid syndrome defined as both persistent positive antiphospholipid antibodies (40 IU or more of anticardiolipin or anti beta2 GPI IgG or IgM, and/or lupus anticoagulant) and a specific clinical setting (thrombotic or obstetrical, apart from RM)
* women with a contraindication or an indication to a treatment by hydroxychloroquine
* Previous exposure > 4 years to chloroquine or hydroxychloroquine
* impossible follow up

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
A live and viable birth | At delivery
  In case of preterm and/or low birth weight, we define the viability by the decision to transfer the newborn to a neonatal intensive care unit

SECONDARY OUTCOMES:
a live and viable birth (for the subgroup analyses) | At delivery
occurrence of pregnancy complications (Recurrent Miscarriage-any other premature termination of pregnancy-placental vascular disease) | Since the beginning of pregnancy up to delivery
gestation time (in weeks of amenorrhea) at delivery, | At delivery up
birth weight (in grams) at delivery | At delivery
survival of the newborn | At 28 days of the newborn
psychomotor development of the child (normal/abnormal) | at 6 months of age
psychomotor development of the child (normal/abnormal) | at 12 months of age
height (in centimeters) | at 6 months of age
height (in centimeters) | at 12 months of age
weight (in grams) | at 6 months of age
weight (in grams) | at 12 months of age
Cranial perimeter (in centimeters) | at 6 months of age
Cranial perimeter (in centimeters) | at 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth PASQUIER, MD, Principal Investigator — EA3878 - University Hospital of Brest
Locations (18):
- France (18):
  - Centre Hospitalier Annecy Genevois, Annecy
  - CH d'Auch, Auch
  - CHU Besançon, Besançon
  - CHRU de Brest, Brest
  - CHU Estaing, Clermont-Ferrand
  - CHRU de Lille, Lille
  - Hôpital Nord - Unité mère-enfant, Marseille
  - CH de Mont de Marsan, Mont-de-Marsan
  - CHU de Nantes, Nantes
  - Hopital Saint Antoine, Paris
  - Hôpital Bichat, Paris
  - Hopital Port Royal Cochin, Paris
  - CHG François Mitterand, Pau
  - Centre hospitalier de Cornouaille, Quimper
  - Hôpital sud de Rennes, Rennes
  - CHU de Saint Etienne - Hôpital Nord, Saint-Etienne
  - Nouvel Hôpital Civil, Strasbourg
  - CH de Bigorre, Tarbes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pasquier E, de Saint-Martin L, Marhic G, Chauleur C, Bohec C, Bretelle F, Lejeune-Saada V, Hannigsberg J, Plu-Bureau G, Cogulet V, Merviel P, Mottier D. Hydroxychloroquine for prevention of recurrent miscarriage: study protocol for a multicentre randomised placebo-controlled trial BBQ study. BMJ Open. 2019 Mar 20;9(3):e025649. doi: 10.1136/bmjopen-2018-025649. PMID 30898821